CLINICAL TRIAL: NCT06644690
Title: The Effect of a Creative Dance-Supported CO-OP Approach on Executive Functions, Attention, Memory, and Dual-Task Performance in Older Adults With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Creative Dance-Supported CO-OP Approach in Older Adults With Mild Cognitive Impairment
Acronym: COOP-DANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Assoc. Prof. Dr., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3ca15029ac154211
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Cognitive Rehabilitation; Mild Cognitive Impairment; Executive Function; Creative Dance; Dual-Task Performance; Older Adults; CO-OP Approach
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: In this parallel-group randomized controlled trial, participants will be assigned to one of two groups. The first group will receive the CO-OP approach combined with creative dance, while the second group will receive only the CO-OP intervention. Both groups will participate in 8-week intervention programs, with sessions held three times a week. The outcomes of interest, such as improvements in executive functions, attention, memory, and dual-task performance, will be compared between the two groups at baseline, post-intervention, and follow-up assessments at 3 and 6 months.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor is blinded to the group assignments to ensure objective evaluation of the study outcomes. Participants, care providers, and investigators are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- CO-OP with Creative Dance (Experimental): Participants in this experimental group will receive the CO-OP (Cognitive Orientation to daily Occupational Performance) approach combined with creative dance interventions. The creative dance component will involve simple, structured movements designed to enhance cognitive and motor functions such as attention, memory, and coordination. The intervention will be administered three times per week for 60-minute sessions over an 8-week period. This group will alternate between CO-OP activities and creative dance exercises, integrating both to improve daily functional performance and cognitive abilities.
  Interventions: Behavioral: CO-OP with Creative Dance
- CO-OP Only (Active Comparator): Participants in this active comparator group will receive the CO-OP (Cognitive Orientation to daily Occupational Performance) approach without any additional creative dance interventions. The CO-OP approach will focus on cognitive and metacognitive strategies to improve daily occupational performance. Sessions will take place three times per week for 60 minutes over an 8-week period. This group will engage in problem-solving and goal-setting activities to enhance functional and cognitive outcomes without the integration of dance or physical movement activities.
  Interventions: Behavioral: CO-OP Only

INTERVENTIONS:
Behavioral: CO-OP with Creative Dance — The CO-OP with Creative Dance intervention integrates the Cognitive Orientation to daily Occupational Performance (CO-OP) approach with structured creative dance sessions. The CO-OP approach focuses on improving cognitive and functional performance through goal-setting, problem-solving, and the use of metacognitive strategies. Creative dance sessions involve simple, rhythmic movements aimed at enhancing motor coordination, memory, and attention. This intervention is administered three times per week for 60 minutes over 8 weeks. The sessions alternate between CO-OP activities and creative dance exercises.
  Arms: 1- CO-OP with Creative Dance
Behavioral: CO-OP Only — The CO-OP Only intervention involves the Cognitive Orientation to daily Occupational Performance (CO-OP) approach, which is designed to improve cognitive and functional performance through structured goal-setting, problem-solving, and metacognitive strategies. Participants engage in activities focused on improving their ability to perform daily tasks by using cognitive tools to develop and execute solutions. The intervention is administered three times per week for 60 minutes over an 8-week period. No additional physical or dance activities are included in this arm.
  Arms: CO-OP Only

SUMMARY:
The goal of this clinical trial is to evaluate if the CO-OP (Cognitive Orientation to daily Occupational Performance) approach, supported by creative dance, can improve cognitive functions in older adults with mild cognitive impairment (MCI). The study focuses on the effects of this intervention on executive functions, attention, memory, and dual-task performance.

The main questions this study aims to answer are:

Does the CO-OP approach with creative dance improve executive functions, attention, and memory more than CO-OP alone? How effective is this intervention in enhancing dual-task performance compared to the standard CO-OP approach?

Participants will:

Engage in either the CO-OP intervention alone or the CO-OP approach combined with creative dance for 8 weeks.

Complete cognitive tasks, participate in creative dance activities, and perform daily tasks during the sessions.

DETAILED DESCRIPTION:
This clinical trial aims to assess the effectiveness of a Cognitive Orientation to daily Occupational Performance (CO-OP) approach, enhanced with creative dance, in older adults with mild cognitive impairment (MCI). The CO-OP method is a cognitive rehabilitation strategy that helps individuals improve occupational performance through goal-setting, problem-solving, and the use of metacognitive strategies. In this study, the CO-OP approach will be integrated with creative dance movements, a form of physical and artistic expression known to stimulate both cognitive and motor functions.

The study will enroll 24 participants between the ages of 65 and 85, diagnosed with MCI according to DSM-5 criteria. Participants will be randomly assigned to two groups:

CO-OP with Creative Dance Group: This group will receive the CO-OP intervention along with creative dance sessions. The creative dance component will consist of simple movements designed to improve motor coordination, memory, and attention, all while fostering social interaction and emotional expression.

CO-OP Only Group: This group will undergo the CO-OP approach alone without any creative dance involvement.

The intervention will last for 8 weeks, with three 60-minute sessions each week. During the sessions, participants in the CO-OP with creative dance group will alternate between cognitive tasks and dance-based activities. The sessions are designed to progressively challenge cognitive and motor skills while ensuring safety and comfort for older adults.

The primary outcome measures include improvements in executive functions, attention, memory, and dual-task performance. Cognitive function will be assessed using standardized neuropsychological tests such as the Trail Making Test Part B (for executive function), Stroop Test (for attention), Rey-Osterrieth Complex Figure Test (for memory), and dual-task assessments combining walking with cognitive tasks. Participants' quality of life will be measured using the SF-36 Health Survey, and depression and social isolation will be evaluated through the Geriatric Depression Scale (GDS) and UCLA Loneliness Scale, respectively.

Secondary measures will focus on the potential emotional and social benefits of integrating creative dance into the CO-OP approach. These will include participant feedback on enjoyment and perceived improvements in social interaction and emotional well-being. The trial will also explore whether the addition of creative dance enhances motivation, engagement, and adherence to the intervention.

Data will be collected at baseline, at the end of the 8-week intervention, and again at 3 and 6 months post-intervention to evaluate both short-term and long-term effects. Statistical analysis will be conducted using repeated measures ANOVA to assess changes over time between groups.

This study is expected to provide insights into how integrating creative dance with the CO-OP approach can potentially offer a more holistic and effective intervention for older adults with MCI, addressing both cognitive and physical domains while also promoting social interaction and emotional health.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 85 years old
* Diagnosis of mild cognitive impairment (MCI) according to DSM-5 criteria
* Ability to participate in physical activities, including creative dance movements
* Willingness to attend all study sessions and follow-up assessments
* Able to give informed consent

Exclusion Criteria:

* Diagnosis of a major neurocognitive disorder (e.g., Alzheimer's disease)
* Presence of severe physical impairments that prevent participation in physical activity
* Current use of medications that significantly affect cognitive function
* Participation in another clinical trial within the past 3 months
* History of significant psychiatric disorders (e.g., major depression, schizophrenia)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Executive Function as Measured by the Trail Making Test Part B | Baseline, immediately after the 8-week intervention, and at 3 and 6 months post-intervention
  The primary outcome is the change in executive function, assessed using the Trail Making Test Part B, from baseline to the end of the 8-week intervention. The test evaluates the participant's ability to switch between tasks, a key component of executive function. Improvements in test scores indicate enhanced cognitive flexibility and task-switching abilities. This outcome is critical for evaluating the impact of the CO-OP approach (with or without creative dance) on executive function in participants with mild cognitive impairment. If you have additional primary measures, they can be included, but typically this would be the focus.

SECONDARY OUTCOMES:
Change in Attention as Measured by the Stroop Test | Baseline, immediately after the 8-week intervention, and at 3 and 6 months post-intervention
  This secondary outcome evaluates changes in attention and cognitive control, assessed using the Stroop Test. The test measures participants' ability to inhibit cognitive interference and focus on relevant stimuli. Improvement in scores from baseline to post-intervention and follow-up points will indicate enhanced attention and cognitive control
Change in Memory Performance as Measured by the Rey-Osterrieth Complex Figure Test | Baseline, immediately after the 8-week intervention, and at 3 and 6 months post-intervention
  This secondary outcome assesses changes in visual memory and organizational skills, using the Rey-Osterrieth Complex Figure Test. Participants' ability to recall and reproduce complex figures will be measured at baseline, post-intervention, and during follow-up assessments at 3 and 6 months. Improvements in scores will indicate enhanced memory function.
Change in Dual-Task Performance as Measured by Walking While Performing a Cognitive Task" | Baseline, immediately after the 8-week intervention, and at 3 and 6 months post-intervention
  This secondary outcome evaluates the participants' ability to perform a motor task (walking) while simultaneously engaging in a cognitive task (such as recalling numbers or words). The assessment will measure the impact of the intervention on dual-task performance, with data collected at baseline, post-intervention, and at 3 and 6 months follow-up. Improvement in dual-task performance will indicate better cognitive-motor integration and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyhun Türkmen, PhD, Principal Investigator — Çankırı Karatekin University
Locations (2):
- Turkey (Türkiye) (2):
  - Çankırı Karatekin University, Faculty of Health Sciences, Çankırı, Not Applicable For Türkiye
  - Ceyhun Türkmen, Çankırı

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhu Y, Gao Y, Guo C, Qi M, Xiao M, Wu H, Ma J, Zhong Q, Ding H, Zhou Q, Ali N, Zhou L, Zhang Q, Wu T, Wang W, Sun C, Thabane L, Zhang L, Wang T. Effect of 3-Month Aerobic Dance on Hippocampal Volume and Cognition in Elderly People With Amnestic Mild Cognitive Impairment: A Randomized Controlled Trial. Front Aging Neurosci. 2022 Mar 10;14:771413. doi: 10.3389/fnagi.2022.771413. eCollection 2022. PMID 35360212
- [Result] Yang HL, Chu H, Kao CC, Miao NF, Chang PC, Tseng P, O'Brien AP, Chou KR. Construction and evaluation of multidomain attention training to improve alertness attention, sustained attention, and visual-spatial attention in older adults with mild cognitive impairment: A randomized controlled trial. Int J Geriatr Psychiatry. 2020 May;35(5):537-546. doi: 10.1002/gps.5269. Epub 2020 Feb 14. PMID 31994767
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Tricco AC, Soobiah C, Berliner S, Ho JM, Ng CH, Ashoor HM, Chen MH, Hemmelgarn B, Straus SE. Efficacy and safety of cognitive enhancers for patients with mild cognitive impairment: a systematic review and meta-analysis. CMAJ. 2013 Nov 5;185(16):1393-401. doi: 10.1503/cmaj.130451. Epub 2013 Sep 16. PMID 24043661
- [Result] Puente AN, Terry DP, Faraco CC, Brown CL, Miller LS. Functional impairment in mild cognitive impairment evidenced using performance-based measurement. J Geriatr Psychiatry Neurol. 2014 Dec;27(4):253-8. doi: 10.1177/0891988714532016. Epub 2014 Apr 24. PMID 24763070
- [Result] Pikouli FA, Moraitou D, Papantoniou G, Sofologi M, Papaliagkas V, Kougioumtzis G, Poptsi E, Tsolaki M. Metacognitive Strategy Training Improves Decision-Making Abilities in Amnestic Mild Cognitive Impairment. J Intell. 2023 Sep 11;11(9):182. doi: 10.3390/jintelligence11090182. PMID 37754911
- [Result] Missiuna C, Mandich AD, Polatajko HJ, Malloy-Miller T. Cognitive orientation to daily occupational performance (CO-OP): part I--theoretical foundations. Phys Occup Ther Pediatr. 2001;20(2-3):69-81. PMID 11345513
- [Result] Lazarou I, Parastatidis T, Tsolaki A, Gkioka M, Karakostas A, Douka S, Tsolaki M. International Ballroom Dancing Against Neurodegeneration: A Randomized Controlled Trial in Greek Community-Dwelling Elders With Mild Cognitive impairment. Am J Alzheimers Dis Other Demen. 2017 Dec;32(8):489-499. doi: 10.1177/1533317517725813. Epub 2017 Aug 25. PMID 28840742
- [Result] Kattenstroth JC, Kalisch T, Holt S, Tegenthoff M, Dinse HR. Six months of dance intervention enhances postural, sensorimotor, and cognitive performance in elderly without affecting cardio-respiratory functions. Front Aging Neurosci. 2013 Feb 26;5:5. doi: 10.3389/fnagi.2013.00005. eCollection 2013. PMID 23447455
- [Result] Frith E, Ryu S, Kang M, Loprinzi PD. Systematic Review of the Proposed Associations between Physical Exercise and Creative Thinking. Eur J Psychol. 2019 Dec 19;15(4):858-877. doi: 10.5964/ejop.v15i4.1773. eCollection 2019 Dec. PMID 33680164
- [Result] Davydow DS, Hough CL, Levine DA, Langa KM, Iwashyna TJ. Functional disability, cognitive impairment, and depression after hospitalization for pneumonia. Am J Med. 2013 Jul;126(7):615-24.e5. doi: 10.1016/j.amjmed.2012.12.006. Epub 2013 Mar 14. PMID 23499326
- [Result] Davies SJ, Gullo HL, Doig E. Efficacy and Feasibility of the CO-OP Approach in Parkinson's Disease: RCT Study Protocol. Can J Occup Ther. 2023 Dec;90(4):363-373. doi: 10.1177/00084174231156287. Epub 2023 Feb 13. PMID 36785891
- [Result] Coelho P, Marmeleira J, Cruz-Ferreira A, Laranjo L, Pereira C, Bravo J. Creative dance associated with traditional Portuguese singing as a strategy for active aging: a comparative cross-sectional study. BMC Public Health. 2022 Mar 29;21(Suppl 2):2334. doi: 10.1186/s12889-022-12978-4. PMID 35351064
- [Result] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Result] Castellote-Caballero Y, Carcelen Fraile MDC, Aibar-Almazan A, Afanador-Restrepo DF, Gonzalez-Martin AM. Effect of combined physical-cognitive training on the functional and cognitive capacity of older people with mild cognitive impairment: a randomized controlled trial. BMC Med. 2024 Jul 8;22(1):281. doi: 10.1186/s12916-024-03469-x. PMID 38972988
- [Result] Casagrande M, Marselli G, Agostini F, Forte G, Favieri F, Guarino A. The complex burden of determining prevalence rates of mild cognitive impairment: A systematic review. Front Psychiatry. 2022 Sep 23;13:960648. doi: 10.3389/fpsyt.2022.960648. eCollection 2022. PMID 36213927
- [Result] Burzynska AZ, Jiao Y, Knecht AM, Fanning J, Awick EA, Chen T, Gothe N, Voss MW, McAuley E, Kramer AF. White Matter Integrity Declined Over 6-Months, but Dance Intervention Improved Integrity of the Fornix of Older Adults. Front Aging Neurosci. 2017 Mar 16;9:59. doi: 10.3389/fnagi.2017.00059. eCollection 2017. PMID 28360853
- [Result] Britten L, Pina I, Nykjaer C, Astill S. Dance on: a mixed-method study into the feasibility and effectiveness of a dance programme to increase physical activity levels and wellbeing in adults and older adults. BMC Geriatr. 2023 Jan 26;23(1):48. doi: 10.1186/s12877-022-03646-8. PMID 36703116
- [Result] Balbim GM, Aguinaga S, Ajilore OA, Bustamante EE, Erickson KI, Lamar M, Marquez DX. The Effects of the BAILAMOSTM Dance Program on Physical Activity Levels and Cognition of Older Latino Adults: A Pilot Study. J Aging Health. 2022 Jan;34(1):25-40. doi: 10.1177/08982643211020996. Epub 2021 May 22. PMID 34027686
- [Result] Appleton E, Maeir T, Kaufman Y, Karni S, Gilboa Y. Cognitive Orientation to daily Occupational Performance (CO-OP) for Older Adults After a Hip Fracture: A Pilot Study. Am J Occup Ther. 2023 Jan 1;77(1):7701205130. doi: 10.5014/ajot.2023.050073. PMID 36779978
- [Result] Altuntas O, Degerli MNO, Temizkan E, Ekici G. Psychometric properties of the Canadian occupational performance measure in older individuals. Turk J Med Sci. 2023 Nov 28;54(1):338-347. doi: 10.55730/1300-0144.5796. eCollection 2024. PMID 38812638